CLINICAL TRIAL: NCT02508753
Title: A Double-Blind, Double-Dummy, Randomized, Moxifloxacin and Placebo Controlled, Four-Way Crossover Study of the Effects of a Single Intravenous Supra-Therapeutic Dose and Single Intravenous Therapeutic Dose of CXA-101/Tazobactam on the QT/QTC Intervals in Healthy Subjects
Brief Title: Safety Study Designed to Study the Effects of Two Different Doses of CXA-101/Tazobactam, a Low Dose and a High Dose, on the QT/QTc Intervals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 7625A-033; CXA-QT-10-02 (Other: Cubist Protocol Number)
Record Dates: First submitted 2010-06-17; First posted 2015-07-27 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: QT/QTc Intervals
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CXA-101/tazobactam therapeutic dose (Experimental)
  Interventions: Drug: CXA-101/tazobactam
- CXA-101/tazobactam supra-therapeutic dose (Experimental)
  Interventions: Drug: CXA-101/tazobactam
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CXA-101/tazobactam — 1000/500 mg single IV dose administered over 60 minutes
  Arms: CXA-101/tazobactam therapeutic dose
Drug: CXA-101/tazobactam — 3000/1500 mg single IV dose administered over 60 minutes
  Arms: CXA-101/tazobactam supra-therapeutic dose
Drug: Moxifloxacin — 400 mg tablet
  Arms: Moxifloxacin
Drug: placebo — single IV dose of a saline solution administered over 60 minutes plus oral over-encapsulated moxifloxacin placebo tablet administered at the start of infusion.
  Arms: Placebo

SUMMARY:
The purpose of the study is look at the possible side effects of two different doses of CXA-101/tazobactam, a low dose and a high dose, on participant's heart.

DETAILED DESCRIPTION:
Some drugs can have effects on the cardiovascular system (hearts and blood vessels) including the QT interval. The QT interval is the time between the contraction and relaxation of the chambers of the heart, called ventricles, which collect and pump blood. The use of some drugs can lead to serious issues such as QT interval prolongation (lengthen) and potentially serious arrhythmias (abnormal heart beat), and sudden death. Therefore, it is important to study effect of medications on the heart.

The drug, Moxifloxacin, will be introduced as a control to be able to compare the effect, if any, that CXA 101/tazobactam might have on participant's heart.Moxifloxacin is an approved antibiotic commonly used to treat common bacterial infections. Moxifloxacin is known to slightly increase the electrical conduction of participant's heart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and/or female, 18-45 years of age who can provide written Informed Consent.
* Body mass index (BMI) between 18-30, inclusive.
* Medically healthy with no clinically significant abnormal screening results (laboratory profiles, medical histories, ECGs, physical exam.
* Voluntarily consent to participate in the study.
* Normal blood pressure (<140 mmHg systolic and <90 mmHg diastolic).
* Normal 12-lead ECG, as defined as:

Consistent sinus rhythm No clinically significant conduction disorders PR interval between 120 and 210 milliseconds (msec), inclusive Heart rate (HR) greater than or equal to 50 beats per minute (bpm) and less than or equal to 100 bpm QRS interval less than or equal to 110 msec QT intervals that can be consistently analyzed (T wave amplitude 2 mm or greater, lack of artifact [noise] and excessive baseline wandering, without any form of bundle branch block).

* QTcF interval less than or equal to 430 msec for males and less than or equal to 450 msec for females.
* Calculated creatinine clearance >80 mL/min. at screening using the Cockcroft-Gault formula.
* If female, subject must have a negative serum pregnancy test at screening and agrees to either be sexually inactive (abstinent) for 14 days prior to screening and throughout the study, or use one of the following acceptable birth control methods:

  1. Intrauterine device (IUD) in place for at least 2 months prior to Day 1 and through study completion; or,
  2. Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; or
  3. Stable hormonal contraceptive (with the same medication, if possible) for at least 3 months prior to Day 1 through one month after completion of study; or
  4. Surgical sterilization (vasectomy) of partner at least 6 months prior to Day 1; or
  5. Naturally postmenopausal for a minimum of 2 consecutive years prior to Day 1; or
  6. Surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to Day 1, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to Day 1).
* If male, subject agrees to use a medically acceptable contraceptive defined as:

  1. Abstain from sexual intercourse through study completion; or
  2. Use a condom with spermicide through study completion; or
  3. Have had a vasectomy at least 6 months prior to Day 1; or
  4. Have a partner who is not of childbearing potential, through study completion.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* History of additional risk factors for Torsade de Pointes (e.g., hypokalemia, family history of long QT Syndrome, family history of Short QT Syndrome, or family history of unexplainable early sudden death).
* History of invasive cancer within the past 5 years (excluding non-melanoma skin cancers).
* History of sensitivity or allergy to the quinolone class of antibiotics, cephalosporin class of antibiotics, or the beta-lactam class of antibiotics.
* History or presence of alcoholism or drug abuse within the past 2 years.
* History of hepatitis B, hepatitis C, Human Immunodeficiency Virus (HIV).
* History of clinically significant syncope.
* History of clinically significant psychiatric illness that would prevent the subject from providing a valid Informed Consent Form (ICF).
* Use of tobacco products within the previous 6 months.
* Donation of blood within 45 days prior to Study Day 1.
* Plasma donation within 30 days prior to Study Day 1.
* Participation in a study of an investigational drug within 30 days prior to the baseline ECG.
* Participation in another clinical trial within 30 days prior to the day of check-in for this study.
* Female and pregnant or lactating.
* Has angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality.
* Positive laboratory results for substances of abuse, cotinine, or alcohol.
* Taken any prescription medication (with the exception of hormonal birth control medications or hormone replacement therapy) within 14 days (or 5 elimination half-lives, whichever is longer) of admission to the unit (Day -2), or have taken any over the counter (OTC) medications, including topical medications, vitamins, herbal or dietary supplements/remedies (e.g., Saint John's Wort or Milk Thistle), within 14 days of admission, or planned concomitant medication while in the study (except for acetaminophen or naproxen, if needed for headache or pain).
* In the opinion of the Investigator, subject would not be able to provide reliable study data or be available for study follow-up.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The change from the pre-dose baseline in the individual subject (subject-specific) correction, QTcI. | Baseline through Day 13
  The primary endpoint is the baseline-adjusted change in the QTcI between time-matched placebo and study drug.
The change from the periodic specific pre-dose baseline of QT/QTcI | Baseline through Day 13
  The primary endpoint is the change from the periodic specific pre-dose baseline of QT/QTcI corrected by QTcI across all dose groups

SECONDARY OUTCOMES:
The change from pre-dose baseline in the QT/QTcI corrected by QTcB and QTcF interval. | Baseline through Day 13
Characterize concentration-response relationship for QT/QTcI | Baseline through Day 13
Provide safety information by the collection of adverse events | Baseline through Day 21
  Collect AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Reserach, Fargo, North Dakota, United States